CLINICAL TRIAL: NCT00809328
Title: A Multicenter, Non-Randomized, Open Label Study Of Azithromycin Intravenous Followed By Oral Administration In Japanese Adult Subjects With Community Acquired Pneumonia (CAP) Requiring Initial Intravenous Therapy
Brief Title: The Study Of Azithromycin Switch Therapy For Treatment Of Community Acquired Pneumonia (CAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661191
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Community Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): Azithromycin switch therapy (switch from intravenous to oral)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — The intravenous formulation 500 mg is administered once daily for 2-5 days; followed by the oral formulation 500 mg will be given once daily to complete a 7 to 10-day course of therapy.

SUMMARY:
Azithromycin has high rates of clinical response and eradication, wide spectrum of activity, so we suppose the development of the azithromycin injectable formulation in Japan would deliver benefit to patients of community acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older patients with CAP.
* Patients who were diagnosed as moderate in severity.

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance to azithromycin, other macrolides, or ketolides.
* Hepatic dysfunction (AST, ALT, total bilirubin > 3 times institutional normal).
* Severe renal dysfunction (creatinine clearance < 30 ml/min).
* Patients who have a history of severe heart diseases (4th -degree of NYHA). Patients who have a congenital or sporadic long QT syndrome, or who are received the drugs with reported QT prolongation.
* Severe underlying disease.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- Japan (34):
  - Pfizer Investigational Site, Seto-shi, Aichi-ken
  - Pfizer Investigational Site, Touon, Ehime
  - Pfizer Investigational Site, Chikushino-shi, Fukuoka
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Koga, Fukuoka
  - Pfizer Investigational Site, Yanagawa, Fukuoka
  - Pfizer Investigational Site, Higashihiroshima, Hiroshima
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Asahikawa, Hokkaido
  - Pfizer Investigational Site, Himejishi, Hyōgo
  - Pfizer Investigational Site, Moriya, Ibaraki
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Takamatsu, Kagawa-ken
  - Pfizer Investigational Site, Kawasaki, Kanagawa
  - Pfizer Investigational Site, Kochi, Kochi
  - Pfizer Investigational Site, Tsu, Mie-ken
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Matsumoto, Nagano
  - Pfizer Investigational Site, Emukae, Kitamatsuura, Nagasaki
  - Pfizer Investigational Site, Isahaya, Nagasaki
  - Pfizer Investigational Site, Nagasaki, Nagasaki
  - Pfizer Investigational Site, Sasebo, Nagasaki
  - Pfizer Investigational Site, Niigata, Niigata
  - Pfizer Investigational Site, Ōita, Oita Prefecture
  - Pfizer Investigational Site, Yufu, Oita Prefecture
  - Pfizer Investigational Site, Kurashiki, Okayama-ken
  - Pfizer Investigational Site, Okinawa, Okinawa
  - Pfizer Investigational Site, Sakai, Osaka
  - Pfizer Investigational Site, Ureshinoshi, Saga-ken
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Meguro-Ku, Tokyo
  - Pfizer Investigational Site, Toshima-ku, Tokyo
  - Pfizer Investigational Site, Yonezawa, Yamagata
  - Pfizer Investigational Site, Shiogama

REFERENCES:
- [Derived] Kohno S, Tateda K, Kadota J, Fujita J, Niki Y, Watanabe A, Nagashima M. Contradiction between in vitro and clinical outcome: intravenous followed by oral azithromycin therapy demonstrated clinical efficacy in macrolide-resistant pneumococcal pneumonia. J Infect Chemother. 2014 Mar;20(3):199-207. doi: 10.1016/j.jiac.2013.10.010. Epub 2013 Dec 11. PMID 24477328
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661191&StudyName=The%20Study%20Of%20Azithromycin%20Switch%20Therapy%20For%20Treatment%20Of%20Community%20Acquired%20Pneumonia%20%28CAP%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: Azithromycin switch therapy (from 500 mg intravenous azithromycin once daily for 2 to 5 days to 500 mg oral azithromycin once daily to complete a total of 7 to 10 days therapy)
Period: Overall Study
Arm/Group | Azithromycin
Started | 102
Completed | 73
Not Completed | 29
Not completed — Lack of Efficacy | 18
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin
Number analyzed (Participants) | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Clinical Response, Data Review Committee Assessment)
Description: Response rate was calculated from the following formula, "the number of participants assessed as effective" over "total participants excluding ones assessed as indeterminate" multiplied by 100.
Time Frame: End of Treatment, Day 15 and Day 29
Population: Clinical per protocol set consisted of all subjects who received at least one dose of the study drug, have no significant violation of protocol, and underwent prescribed evaluations during the observation period. No imputation was used for missing data. "n " in the measured values means total participants excluding ones assessed as indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 73
percentage of participants
  End of Treatment (n=73) | 86.3 [76.2 to 93.2]
  Day 15 (Primary analysis ) (n=71) | 84.5 [74.0 to 92.0]
  Day 29 (n=70) | 82.9 [72.0 to 90.8]

2. Secondary Outcome: Response Rate (Clinical Response, Investigator Assessment)
Description: as for outcome 1
Time Frame: End of Treatment, Day 15 and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 73
percentage of participants
  End of Treatment (n=73) | 80.8 [69.9 to 89.1]
  Day 15 (n=62) | 98.4 [91.3 to 100.0]
  Day 29 (n=61) | 95.1 [86.3 to 99.0]

3. Secondary Outcome: The Tendency Toward Clinical Improvement (Investigator Assessment)
Description: The number of participants who showed tendency toward clinical improvement based on the assessment of temperature, white blood cell count, C-reactive protein, clinical symptoms on Day 3, and was determined to continue the treatment.
Time Frame: Day 3
Population: Clinical per protocol set consisted of all subjects who received at least one dose of the study drug, have no significant violation of protocol, and underwent prescribed evaluations during the observation period. No imputation was used for missing data.
Measure: Number; unit: participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 73
participants | 68

4. Secondary Outcome: Eradication Rate (Bacteriological Response, Data Review Committee Assessment)
Description: Eradication Rate was calculated from the following formula, "the number of participants assessed as eradication , presumed eradication or microbial substitution" over "total participants excluding ones assessed as indeterminate" multiplied by 100
Time Frame: Day 3, End of Treatment, Day 15 and Day 29
Population: Bacteriologic per protocol set consisted of all subjects in the clinical per protocol set in whom bacterial pathogens were identified at baseline. No imputation was used for missing data. "n " in the measured values was the total participants EXCLUDING ones assessed as indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 33
percentage of participants
  Day 3 (n=28) | 71.4 [51.3 to 86.8]
  End of Treatment (n=31) | 80.6 [62.5 to 92.5]
  Day 15 (n=30) | 83.3 [65.3 to 94.4]
  Day 29 (n=30) | 83.3 [65.3 to 94.4]

5. Secondary Outcome: Eradication Rate (Bacteriological Response, Investigator Assessment)
Description: as for outcome 4
Time Frame: Day 3, End of Treatment, Day 15 and Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentageof participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 33
percentageof participants
  Day 3 (n=27) | 74.1 [53.7 to 88.9]
  End of Treatment (n=29) | 86.2 [68.3 to 96.1]
  Day 15 (n=25) | 100.0 [86.3 to 100.0]
  Day 29 (n=25) | 100.0 [86.3 to 100.0]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Azithromycin
Serious Adverse Events (participants affected / at risk) | 8/102
Other Adverse Events (participants affected / at risk) | 33/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=102)
Cardiac failure congestive (Cardiac disorders) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Prothrombin time prolonged (Investigations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=102)
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 15
Injection site erythema (General disorders) | 3
Injection site pain (General disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.